CLINICAL TRIAL: NCT00880971
Title: Post-Operative Radiation Therapy for Patients With pⅢA-N2 Non-Small Cell Lung Cancer After Complete Resection and Adjuvant Chemotherapy: A Prospective Randomized Phase Ⅲ Study
Brief Title: Postoperative Radiotherapy for Patients With IIIA (N2) Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Chairman of Thoracic Group, Clinical Professor, Radiation Oncology Department, Cancer Hospital&Institute, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-015
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Thoracic Neoplasms; Non-small Cell Lung Cancer
Keywords: Lung; Carcinoma; radiotherapy; Surgery
MeSH Terms: conditions — Thoracic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PORT (Experimental): Patients undergo thoracic radiotherapy using 3D-CRT or IMRT (50 Gy, 2 Gy once daily over 5 weeks) after postoperative chemotherapy.
  Interventions: Radiation: Postoperative 3D-CRT or IMRT
- Non-PORT (No Intervention): Patients undergo postoperative chemotherapy.

INTERVENTIONS:
Radiation: Postoperative 3D-CRT or IMRT — Postoperative radiotherapy using 3D-CRT or IMRT techniques, 2 Gy per fraction, total 25 fractions (50Gy) over 5 weeks.
  Other Names: Postoperative radiotherapy
  Arms: PORT

SUMMARY:
Several important international randomized trials have shown that postoperative chemotherapy contributed to the improvement on 5 year survival rate by about 4% for patients with non-small cell lung cancer (NSCLC) after complete resection. But the overall survival rate was relatively low and the local recurrence was still the dominant failure pattern for stage IIIA (N2) disease even these patients received the postoperative chemotherapy. Several meta-analyses have shown that postoperative radiotherapy (PORT) has no effect on the survival improvement for patients with NSCLC after complete resection. However, sub-group analysis based on the same dataset of these meta-analyses showed that the PORT with conventional radiotherapy might be beneficial for stage IIIA (N2) disease. The 3D conform radiotherapy (3D-CRT) and intensity modified radiotherapy (IMRT) can increase the radiation dose to the target volume while decreasing the dose to risk organs comparing with the conventional radiotherapy. So it is expected that PORT using 3D-CRT or IMRT after postoperative chemotherapy will improve the local control and survival for stage IIIA (N2) NSCLC. Here, the investigators designed a phase III randomized trial to compare the 3-year disease free survival (DFS) and overall survival (OS) rates in patients with completely resected stage IIIA (N2) NSCLC who receive adjuvant chemotherapy alone or adjuvant chemotherapy plus PORT.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: To determine whether administering adjuvant chemotherapy (four cycles of platinum-based doublet regimen) plus PORT (50 Gy, 2 Gy once daily over 5 weeks) will improve 3-year DFS compared with adjuvant chemotherapy alone in patients with completely resected stage IIIA (N2) NSCLC.

Secondary: To compare treatment-related toxic effects, 3-year OS, failure-free survival, and the patterns of failure.

OUTLINE: Eligible patients were randomized equally, using simple randomization, to either PORT or observation group.

Arm I: Patients undergo PORT using 3D-CRT or IMRT (50 Gy, 2 Gy once daily over 5 weeks) after adjuvant chemotherapy.

Arm II: Patients undergo adjuvant chemotherapy.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Completely resected disease by lobectomy, bilobectomy. Complete dissection of lymph nodes at levels 4, 7, and 10 in case of right-sided thoracotomy and at levels 4 (if accessible), 5, 6, 7, and 10 in case of left-sided thoracotomy.
* Histologically N2 disease after surgery. Negative margins
* Has undergone chemotherapy of four cycles of platinum-based doublet regimen and no recurrence and metastasis

Exclusion Criteria:

* Pregnant or nursing
* ECOG performance status > 1
* Post-operative FEV_1 < 1 L (or < 35% theoretical value, PO_2 < 70 mm Hg, and PCO_2 > 45 mm Hg)
* Severe cardiac disease within the past 6 months, including the following: Arrhythmia, Congestive heart failure, Infarction, Pacemaker
* Severe pulmonary disease within the past 6 months
* Other prior or concurrent neoplasm, except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Severe or uncontrolled systemic disease
* Familial, social, geographic, or psychological conditions that would preclude study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2009-02-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
DFS | 3 years
  Disease free survival measures in months.

SECONDARY OUTCOMES:
OS | 3 years
  Overall survival measures in months.
LRFS | 3 years
  Loco-regional recurrence free survival measures in months.
DMFS | 3 years
  Distant metastasis free survival measures in months.
Failure Patterns | 3 years
  Loco-regional recurrence (LR) and Distant metastasis (DM)
Toxicity of thoracic radiotherapy | 6 months
  CTC AE 3.0 is used to evaluate the toxicities, including radiation esophagitis (RE) and pneumonitis (RP).

CONTACTS AND LOCATIONS:
Overall Officials: Luhua Wang, MD, Principal Investigator — Cancer Hosiptal, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hosiptal, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Chemotherapy in non-small cell lung cancer: a meta-analysis using updated data on individual patients from 52 randomised clinical trials. Non-small Cell Lung Cancer Collaborative Group. BMJ. 1995 Oct 7;311(7010):899-909. PMID 7580546
- [Background] Postoperative radiotherapy in non-small-cell lung cancer: systematic review and meta-analysis of individual patient data from nine randomised controlled trials. PORT Meta-analysis Trialists Group. Lancet. 1998 Jul 25;352(9124):257-63. PMID 9690404
- [Background] Keller SM, Adak S, Wagner H, Herskovic A, Komaki R, Brooks BJ, Perry MC, Livingston RB, Johnson DH. A randomized trial of postoperative adjuvant therapy in patients with completely resected stage II or IIIA non-small-cell lung cancer. Eastern Cooperative Oncology Group. N Engl J Med. 2000 Oct 26;343(17):1217-22. doi: 10.1056/NEJM200010263431703. PMID 11071672
- [Background] Lally BE, Zelterman D, Colasanto JM, Haffty BG, Detterbeck FC, Wilson LD. Postoperative radiotherapy for stage II or III non-small-cell lung cancer using the surveillance, epidemiology, and end results database. J Clin Oncol. 2006 Jul 1;24(19):2998-3006. doi: 10.1200/JCO.2005.04.6110. Epub 2006 Jun 12. PMID 16769986
- [Background] Machtay M, Lee JH, Shrager JB, Kaiser LR, Glatstein E. Risk of death from intercurrent disease is not excessively increased by modern postoperative radiotherapy for high-risk resected non-small-cell lung carcinoma. J Clin Oncol. 2001 Oct 1;19(19):3912-7. doi: 10.1200/JCO.2001.19.19.3912. PMID 11579111
- [Background] Matsuguma H, Nakahara R, Ishikawa Y, Suzuki H, Inoue K, Katano S, Yokoi K. Postoperative radiotherapy for patients with completely resected pathological stage IIIA-N2 non-small cell lung cancer: focusing on an effect of the number of mediastinal lymph node stations involved. Interact Cardiovasc Thorac Surg. 2008 Aug;7(4):573-7. doi: 10.1510/icvts.2007.174342. Epub 2008 Apr 15. PMID 18413349
- [Background] Douillard JY, Rosell R, De Lena M, Riggi M, Hurteloup P, Mahe MA; Adjuvant Navelbine International Trialist Association. Impact of postoperative radiation therapy on survival in patients with complete resection and stage I, II, or IIIA non-small-cell lung cancer treated with adjuvant chemotherapy: the adjuvant Navelbine International Trialist Association (ANITA) Randomized Trial. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):695-701. doi: 10.1016/j.ijrobp.2008.01.044. Epub 2008 Apr 24. PMID 18439766
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] Ng R, Hasan B, Mittmann N, Florescu M, Shepherd FA, Ding K, Butts CA, Cormier Y, Darling G, Goss GD, Inculet R, Seymour L, Winton TL, Evans WK, Leighl NB; Working Group on Economic Analysis; Lung Disease Site Group; National Cancer Institute of Canada Clinical Trials Group. Economic analysis of NCIC CTG JBR.10: a randomized trial of adjuvant vinorelbine plus cisplatin compared with observation in early stage non-small-cell lung cancer--a report of the Working Group on Economic Analysis, and the Lung Disease Site Group, National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 Jun 1;25(16):2256-61. doi: 10.1200/JCO.2006.09.4342. PMID 17538170
- [Background] Dunant A, Pignon JP, Le Chevalier T. Adjuvant chemotherapy for non-small cell lung cancer: contribution of the International Adjuvant Lung Trial. Clin Cancer Res. 2005 Jul 1;11(13 Pt 2):5017s-5021s. doi: 10.1158/1078-0432.CCR-05-9006. PMID 16000606
- [Derived] Men Y, Bao Y, Bi N, Zhou Z, Liang J, Lv J, Feng Q, Xiao Z, Wang Y, Li J, Wang J, Gao S, He J, Hui Z, Wang L. Long-term outcomes of postoperative radiotherapy for patients with pIIIA-N2 non-small-cell lung cancer after complete resection and adjuvant chemotherapy (PORT-C): a single-centre, randomized, phase 3 trial. EClinicalMedicine. 2025 Oct 16;89:103503. doi: 10.1016/j.eclinm.2025.103503. eCollection 2025 Nov. PMID 41146922
- [Derived] Hui Z, Men Y, Hu C, Kang J, Sun X, Bi N, Zhou Z, Liang J, Lv J, Feng Q, Xiao Z, Chen D, Wang Y, Li J, Wang J, Gao S, Wang L, He J. Effect of Postoperative Radiotherapy for Patients With pIIIA-N2 Non-Small Cell Lung Cancer After Complete Resection and Adjuvant Chemotherapy: The Phase 3 PORT-C Randomized Clinical Trial. JAMA Oncol. 2021 Aug 1;7(8):1178-1185. doi: 10.1001/jamaoncol.2021.1910. PMID 34165501
- [Derived] Wang J, Hui Z, Men Y, Kang J, Sun X, Deng L, Zhai Y, Wang W, Bi N, Liang J, Lv J, Zhou Z, Feng Q, Xiao Z, Chen D, Wang L, Zhao J. Systemic Inflammation-Immune Status Predicts Survival in Stage III-N2 Non-Small Cell Lung Cancer. Ann Thorac Surg. 2019 Dec;108(6):1701-1709. doi: 10.1016/j.athoracsur.2019.06.035. Epub 2019 Aug 7. PMID 31400325